CLINICAL TRIAL: NCT04480255
Title: NICU2HOME+: Supporting Illinois Families of Premature Infants With Smartphone Technology
Brief Title: NICU2HOME+: Supporting Illinois Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Craig Garfield, Professor of Pediatrics; and Attending physician and neonatal hospitalist at the Lurie Children's Hospital of Chicago where he is the Director of Research for the Division, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00212196
Record Dates: First submitted 2020-07-08; First posted 2020-07-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Premature Birth; NICU; Premature; Infant
Keywords: Premature Infant; NICU; Premature Birth; Smartphone App; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Standard of Care (Active Comparator): Parents of infants born from date July 2020-December 2020
  Interventions: Other: Group 1: Standard of Care
- Group 2: NICU2HOME+ app (Active Comparator): Parents of infants born from mid Jan 2021-May2021
  Interventions: Other: Group 2: NICU2HOME+ app

INTERVENTIONS:
Other: Group 1: Standard of Care — Those who are in Group 1 will receive the usual care which includes:
  1. a welcome packet from the nursing staff
  2. access to their infant's medical team including doctors and nurse
  3. opportunities to ask any questions and understand the care their baby is receiving through participation in daily work rounds or through setting up family meetings with the medical team.
  Arms: Group 1: Standard of Care
Other: Group 2: NICU2HOME+ app — In addition to the usual care made available to Group 1 as described above, Group 2 parents will receive the smartphone app. Group 2 parents will be asked to download the NICU2HOME app.
  Arms: Group 2: NICU2HOME+ app

SUMMARY:
The purpose of this project is to provide a stepwise, methodical approach to developing and testing the ability of Neonatal Intensive Care Unit 2 Home (NICU2HOME+) to support diverse Illinois families of premature infants during and after their Neonatal Intensive Care Unit (NICU) stays in an effort to address health equity, improve parenting, and reduce costs. There are 3 objectives of the study: 1) Identify and assess the requirements for expansion of NICU2HOME+, a suite of mobile patient education and engagement applications with Electronic Medical Record (EMR) integration that is culturally appropriate and customized to the needs of a diverse population of patients and families to 3 additional level III Illinois NICUS; 2) develop and deploy NICU2HOME+ to these 3 additional NICUs; and 3)determine if it is effective in: a) addressing health equity issues, b) improving parenting self-efficacy and satisfaction, and c) improving NICU outcomes such as a reduced length of stay and lower readmission rates that result in lower healthcare costs.

All research recruitment and participation will take place in the following spaces:

1. Northwestern Medicine's Central DuPage Hospital (25 N.Winfield Rd., Winfield, IL)- NICU, Postpartum, and Research Offices
2. Northwest Community Hospital (800 W. Central Rd., Arlington Heights, IL)- NICU,Postpartum, and Research Offices
3. Rush University Medical Center (Chicago, IL)- NICU, Postpartum, and Research Offices

DETAILED DESCRIPTION:
The investigators propose to address the goals of the Affordability Cures Initiative and promote health equity by developing NICU2HOME+, a smartphone app designed to support NICU parents in a culturally appropriate manner in community level III NICUs in Illinois and to include EMR integration. Mobile technology such as NICU2HOME+ offers an innovative way to reduce costs in two ways. First, parents who are better informed and supported, who feel more confident and competent in caring for their premature infants, may be more prepared for an earlier discharge. Second, cost savings may be realized after discharge, if better educated and more competent parents are less likely to inappropriately visit the ER or their infant's physicians as they know what to expect and can provide better, more competent care to their baby. At its center, NICU2HOME+is able to achieve four "rights" of adaptive personalization and parent-centric care: delivering the "right" information at the "right" time to the "right" person via the "right" medium. The ultimate goal of this proposal, therefore, is to develop a scalable, evidence-based.

Participants will be divided into two research groups based on when their infant was born. The first group, parents of infants born between June 15th and December 31st 2020, will receive the standard care provided in the NICU. The second group of participants, those with infants born between January 1 and July 31 2021, will also receive the NICU standard care and additionally be asked to use a smartphone app related to NICU and at-home care. Participation in the second groups requires ownership of a smartphone and the ability to use a smartphone app.

If the participant has been assigned to the first group, the investigators would like both parents to participate in the study independently and therefore complete individual consent forms. However, the investigators recognize not all families will have two parents that are interested or able to participate and ultimately participation from some families will include only one parent.

As part of the study, participants will be asked to complete four surveys. They will be administered at the time of admission, infant's discharge from the NICU, fourteen days after discharge and thirty days after discharge. For those families who have a longer stay in the NICU, the investigators will ask parents to complete two additional surveys; one 30 days after admission and one 60 days after admission.Each survey will take approximately five to ten minutes to complete. The main benefit of participation is that this research that may help improve the NICU experience for other families in the future. The primary risk of participation is the potential loss of confidentiality, but strict measures are in place to minimize the chance of this happening.

In addition, if participants agree to the option at the end of this Consent Form, participants may or may not be invited to participate in a separate research interview to take place during the participants NICU stay, around the time of the infant's discharge from the hospital, or within a year of the transition to home. These optional, voluntary interviews will be conducted at a time, location and method (phone or in-person) agreed upon by the parent. All interviews will be conducted with our research staff with experience interviewing parents of NICU graduates. While the investigators encourage both parents to participate in order to hear about differences in experiences, one or both parents can ultimately participate. The purpose of the research interview is to better understand participants' experience in the NICU and at home as the parent of a premature infant.

Participants will be divided into two research groups based on when their infant was born. The first group, parents of infants born between July 15th and December 31st 2020, will receive the standard care provided in the NICU. The second group of participants, those with infants born between January 1 and July 31 2021, will also receive the NICU standard care and additionally be asked to use a smartphone app related to NICU and at-home care. Participation in the second groups requires ownership of a smartphone and the ability to use a smartphone app.

If a participants are assigned to the first or second groups, the investigators would like both parents to participate in the study independently and therefore complete individual consent forms. However, the investigators recognize not all families will have two parents that are interested or able to participate and ultimately participation from some families will include only one parent.

As part of the study, participants will be asked to complete four surveys. They will be administered at the time of admission, infant's discharge from the NICU, fourteen days after discharge and thirty days after discharge. For those families who have a longer stay in the NICU, the investigators will ask parents to complete two additional surveys; one 30 days after admission and one 60 days after admission. Each survey will take approximately five to ten minutes to complete. The main benefit of participation is that this research that may help improve the NICU experience for other families in the future. The primary risk of participation is the potential loss of confidentiality, but strict measures are in place to minimize the chance of this happening.

In addition, if participants agree to the option at the end of this Consent Form, participants may or may not be invited to participate in a separate research interview to take place during the participants' NICU stay, around the time of the participants' infant's discharge from the hospital, or within a year of the participants transition home. These optional, voluntary interviews will be conducted at a time, location and method (phone or in-person) agreed upon by the parent. All interviews will be conducted with our research staff with experience interviewing parents of NICU graduates. While the investigators encourage both parents to participate in order to hear about differences in experiences, one or both parents can ultimately participate. The purpose of the research interview is to better understand the participants' experience in the NICU and at home as the parent of a premature infant.

Optional Interview:

In addition to the intervention study, optional qualitative interviews will be conducted with participants using a maximum variability approach. Interviews will focus on the following:

* Their overall experience of using the app
* Educational Content
* Relationship/communication through app with extended family/friends
* Readiness for discharge
* Empowerment, ability to communicate better with doctors and nurses, and being able to participate in child health care confidently
* Being ready to go home and did the app help
* Information, communication and support needs across the NICU stay, discharge and beyond

This voluntary interview will be described to parents at the time of consent. To maintain confidentiality all subjects will be given a unique study code (PIN) and all information collected for app development will be linked to that number, not to any other identifier. All documents that include identifiers will be stored in a locked, secure location that only key authorized study personnel (e.g. PI, research team members) will have access to.

The interviews will be audio recorded. The recordings will be given an Identification (ID) number and kept in locked cabinets and on secure computers. The audio recordings will be transcribed and kept on password protected computers. (There will be no personal identifiers (such as names) in the transcribed documents.) After the recordings are transcribed, the audio files will be erased.

Only the people listed on the Authorized Research Personnel list will have access to the data. All paper data will be kept in locked files and rooms. Electronic data will be kept in on password- encrypted computers and files with identifying information will be individually password protected. Names and contact information will be stored only for the purpose of contacting participants. This information will be stored separately from study data and the two will only be linked by a study ID, kept in a password protected document. Upon completion of data collection all name and contact information as will be destroyed by file deletion. All data collected for this study will be kept in a locked, secure location and anything that can be destroyed (deleted, shredded, etc.) after it has been coded, will be.

ELIGIBILITY:
Inclusion Criteria:

* Parents (including single parents) of premature infants (<35 weeks) admitted to Central Dupage Hospital (CDH), Northwest Community Hospital (NCH), and Rush University Medical Center (RUSH)
* Infants born prematurely with a gestational age of <35 weeks
* Minimum stay in NICU of 7 days
* Competent in English or Spanish (i.e. to fully understand the questions asked in the surveys)
* Smartphone owner

Exclusion Criteria:

* Non-adults unable to consent/Cognitively Impaired
* Prisoners or other detained individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Mobile Application Outcome 1 | 2-3 months
  The primary outcome measure understand how the smartphone application improves patient/parent experiences in the NICU. This will be measured through a survey.
Mobile Application Outcome 2 | 2-3 months
  The primary outcome measure will addressing the association of the smartphone application with parenting self-efficacy to improve infants' and parents' health outcomes. This will be measured through a survey.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 2-3 months
  Patient anxiety will be measured through a survey. The response options range from 1 to 4 (Almost never, Sometimes, Often, and Almost always)
Parenting Sense of Competence Scale (PSOC) | 2-3 months
  Self-efficacy will be measured through a survey. The response options range from 1 to 6 (Strongly Disagree to Strongly Agree)
Edinburgh Postnatal Depression Scale (EPDS) | 2-3 months
  Depression will be measured through a survey. The response options range from 0 (for example, no, not at all or no, never again) to 3 (for example, yes, most of the time or yes, very often). The total score ranges from 0 to 30, where higher values indicate more severe symptoms of depression.
Press Ganey Questionnaire (PG) | 2-3 months
  Measures all aspects of patient satisfaction during hospital stay.
Healthcare encounters (HE) | 2-3 months
  Patient satisfaction of healthcare provider's will be measured through survey.
Readmission rate (RR) | 2-3 months
  Readmission rates will be measured through a survey.
User Version of the Mobile Application Rating Scale (uMARS) | 2-3 months
  Quality and reliability of mobile application will be measured through a survey. All items are rated on a 5-point scale from "1. Inadequate" to "5. Excellent"
Perinatal PTSD Questionnaire - Modified (PPQ-M) | 2-3 months
  Perinatal Post-Traumatic Stress Disorder (PTSD) will be measured through a survey.
Coronavirus disease 2019 (COVID-19) Impact Scale | 2-3 months
  Given the uncertainty of the global pandemic, we measuring if COVID will have an impact on the use of the mobile application. This scale is measured on a scale from 1-4 (No Change to Severe), with higher scores mean a worse outcome.
Perceived Stress Scale (PSS) | 2-3 months
  Stress will be measured through a survey. The response options range from 1 to 4 (Never Almost; Never Sometimes; Fairly Often; Very Often). The total score ranges from 0 to 16, where higher values indicate more severe symptoms of stress.
MOS- Social Support Scale (MOS) | 2-3 months
  Social Support will be measured through a survey. The response options range from 1 to 5 (None of the time - All of the time). The survey consists of four separate social support subscales and an overall functional social support index. A higher score for an individual scale or for the overall support index indicates more support.
Health Behavior (HB) | 2-3 months
  Health behavior questions relating to physical health, mental health, stress, breastfeeding, and reproductive health will be measured through a survey.
Centers for Disease Control (CDC) - Hear Her Campaign | 2-3 months
  Questions surrounding maternal mortality and morbidity will be asked through a survey.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Santiago, MA, Study Director — Northwestern University
Locations (3):
- United States (3):
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Centra Dupage Hospital, Winfield, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Understanding Premature Birth and Assuring Healthy Outcomes; Behrman RE, Butler AS, editors. Preterm Birth: Causes, Consequences, and Prevention. Washington (DC): National Academies Press (US); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK11362/ PMID 20669423
- [Background] Garfield CF, Lee Y, Kim HN. Paternal and maternal concerns for their very low-birth-weight infants transitioning from the NICU to home. J Perinat Neonatal Nurs. 2014 Oct-Dec;28(4):305-12. doi: 10.1097/JPN.0000000000000021. PMID 24927295
- [Background] Braveman P. What is health equity: and how does a life-course approach take us further toward it? Matern Child Health J. 2014 Feb;18(2):366-72. doi: 10.1007/s10995-013-1226-9. PMID 23397099
- [Background] Blumenshine P, Egerter S, Barclay CJ, Cubbin C, Braveman PA. Socioeconomic disparities in adverse birth outcomes: a systematic review. Am J Prev Med. 2010 Sep;39(3):263-72. doi: 10.1016/j.amepre.2010.05.012. PMID 20709259
- [Background] MacDorman MF. Race and ethnic disparities in fetal mortality, preterm birth, and infant mortality in the United States: an overview. Semin Perinatol. 2011 Aug;35(4):200-8. doi: 10.1053/j.semperi.2011.02.017. PMID 21798400
- [Background] Pew Research Center: Internet Science & Technology. Mobile technology fact sheet. 2018; http://www.pewinternet.org/fact-sheet/mobile/. Accessed January 14, 2019, 2015.
- [Background] Anderson-Lewis C, Darville G, Mercado RE, Howell S, Di Maggio S. mHealth Technology Use and Implications in Historically Underserved and Minority Populations in the United States: Systematic Literature Review. JMIR Mhealth Uhealth. 2018 Jun 18;6(6):e128. doi: 10.2196/mhealth.8383. PMID 29914860
- [Background] Anoshiravani A, Gaskin G, Kopetsky E, Sandborg C, Longhurst CA. Implementing an Interoperable Personal Health Record in Pediatrics: Lessons Learned at an Academic Children's Hospital. J Particip Med. 2011 Jul 10;3:e30. PMID 21853160
- [Background] Cooper LG, Gooding JS, Gallagher J, Sternesky L, Ledsky R, Berns SD. Impact of a family-centered care initiative on NICU care, staff and families. J Perinatol. 2007 Dec;27 Suppl 2:S32-7. doi: 10.1038/sj.jp.7211840. PMID 18034178
- [Background] De Rouck S, Leys M. Information needs of parents of children admitted to a neonatal intensive care unit: a review of the literature (1990-2008). Patient Educ Couns. 2009 Aug;76(2):159-73. doi: 10.1016/j.pec.2009.01.014. Epub 2009 Mar 24. PMID 19321288
- [Background] Escobar GJ, Joffe S, Gardner MN, Armstrong MA, Folck BF, Carpenter DM. Rehospitalization in the first two weeks after discharge from the neonatal intensive care unit. Pediatrics. 1999 Jul;104(1):e2. doi: 10.1542/peds.104.1.e2. PMID 10390288
- [Background] Garfield CF, Lee YS, Kim HN, Rutsohn J, Kahn JY, Mustanski B, Mohr DC. Supporting Parents of Premature Infants Transitioning from the NICU to Home: A Pilot Randomized Control Trial of a Smartphone Application. Internet Interv. 2016 May;4(Pt 2):131-137. doi: 10.1016/j.invent.2016.05.004. Epub 2016 Jun 4. PMID 27990350
- [Background] Kim HN, Garfield C, Lee YS. Paternal and maternal information and communication technology usage as their very low birth weight infants transition home from the NICU. Int J Hum Comput Interact. 2015;31(1):44-54.
- [Background] Lee Y, Garfield C, Massey N, Chaysinh S, Hassan S. NICU-2-home: Supporting the transition to home from the neonatal intensive care unit using a mobile application. Conference on Human Factors in Computing Systems; May 7 - 11,
- [Background] Gilmore L, Cuskelly M. Factor structure of the Parenting Sense of Competence scale using a normative sample. Child Care Health Dev. 2009 Jan;35(1):48-55. doi: 10.1111/j.1365-2214.2008.00867.x. Epub 2008 Oct 22. PMID 18991983

DOCUMENTS (1):
  • Informed Consent Form (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04480255/ICF_000.pdf